CLINICAL TRIAL: NCT03259672
Title: Influence of Sevoflurane and Desflurane on Postoperative Sore Throat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SevoDesPOST
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Hip Arthroplasty
Keywords: intubation; pharyngitis; remifentanil
MeSH Terms: conditions — Pharyngitis | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Active Comparator)
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental)
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane was used as a maintenance anesthetic agent.
  Arms: Sevoflurane
Drug: Desflurane — Desflurane was used as a maintenance anesthetic agent.
  Arms: Desflurane

SUMMARY:
This investigation is planned to compare the incidence and severity of postoperative sore throat according to the use of sevoflurane or desflurane.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients scheduled for general anesthesia with endotracheal intubation

Exclusion Criteria:

* Difficult airway
* Friable teeth
* Rapid sequence induction
* Recent sore throat
* Recent upper respiratory infection
* Asthma
* Chronic obstructive pulmonary disease
* Chronic cough
* Arrhythmia
* Coronary disease
* Heart failure
* Pregnancy
* Allergy to sevoflurane
* Allergy to desflurane
* Fever after halogenated anesthetics
* Jaundice after halogenated anesthetics
* Malignant hyperthremia
* Allergy to remifentanil
* Friable teeth
* History of head and neck surgery
* Multiple intubation attempts
* Regional anesthetic agents
* Gastric tube
* Dexamethasone
* Severe hypovolemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative sore throat | At 24 hr

SECONDARY OUTCOMES:
Number of participants with postoperative sore throat | At 0, 2, 4 and 24 hr
Number of participants with postoperative hoarseness | At 0, 2, 4 and 24 hr
Number of participants with postoperative cough | At 0, 2, 4 and 24 hr
Number of participants with postoperative nausea | At 0, 2, 4 and 24 hr
Number of participants with postoperative vomiting | At 0, 2, 4 and 24 hr
Number of participants with additional pain medication | At 0, 2, 4 and 24 hr
Visual analogue scale of postoperative pain | At 0, 2, 4 and 24 hr
Number of participants with shivering | At 0, 2, 4 and 24 hr
Requirements of analgesics | At 0, 2, 4 and 24 hr